CLINICAL TRIAL: NCT00761787
Title: Cardiac Allograft Rejection Gene Expression Observational (CARGO) II STUDY
Acronym: CARGOII
Status: Completed | Type: Observational
Sponsor: XDx (Industry)
Responsible Party: Helen Baron, MD Associate Medical Director, XDx, Inc.
Other Study IDs: CARGO II
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Graft Rejection; Heart Disease
Keywords: allograft; rejection; biopsy; gene; expression; cardiology; heart; transplant
MeSH Terms: conditions — Heart Diseases; Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood whole blood white blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Heart transplanted subjects.

SUMMARY:
The Cardiac Allograft Rejection Gene Expression Observational (CARGO) II Study is designed to provide independent evidence of the clinical performance of the non-invasive AlloMap test. Sensitive detection of cardiac allograft rejection and dysfunction is the basis for successful recipient management. The CARGO II Study will assess the correlation between the presence or absence of acute cellular rejection as determined by examination of endomyocardial biopsy specimens with results from the AlloMap Test. Of 17 participating transplant centers, 4 are in North America and 13 are in Europe.

ELIGIBILITY:
Inclusion Criteria:

* New and existing allograft recipients
* All patients (age ≥ 18years) receiving post-transplant care at the enrolling centers

Exclusion Criteria:

* Concurrent enrollment in a double-blind drug trial (immunosuppressive drugs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New and existing cardiac allograft recipients.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2005-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Acute Cellular Rejection(ACR)grades - ACR ISHLT Grades will be determined by centralized pathology reading. The associated AlloMap Test score will be correlated to the biopsy reading. | Scheduled clinic visit

SECONDARY OUTCOMES:
Evaluation of the AlloMap Test and novel gene expression algorithm in guiding management of steroids and calcineurin inhibitors based on the algorithm's capacity to predict future cellular rejection and future graft dysfunction. | more than 2 months following date of transplant
Assessment of clinical utility of the AlloMap Test and novel gene expression algorithms in diagnosis and prediction of humoral rejection. | >2 months after date of transplant

CONTACTS AND LOCATIONS:
Locations (17):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Texas Heart Institute, Houston, Texas
- Austria (2):
  - Medizinische Universität Innsbruck, Klinische Abteilung für Herzchirurgie, Anichstrasse 35, Innsbruck
  - Medical University of Vienna (Medizinische Universität Wien), Währinger Gürtel 18-20, Vienna
- UZ Gasthuisberg, Herestraat 49, Leuven, Belgium
- Toronto General Hospital, Toronto, Ontario, Canada
- Hospital La Pitie, 47 Bd de L, Paris, France
- Germany (4):
  - Herz- und Diabeteszentrum NRW, Georgstraße 11, Bad Oeynhausen
  - Medizinische Hochschule Hannover, Hanover, Carl-Neuberg-Str. 1
  - UKM - Medizinische Klinik und Poliklinik C (Kardiologie und Angiologie), Albert-Schweitzer-Str. 33, Münster
  - Deutsches Herzzentrum Berlin, Augustenburger Platz, State of Berlin
- Ospedali Riuniti di Bergamo, Largo Barozzi 1, Bergamo, Italy
- Silesian Center for Heart Disease, Ul. Szpitalna 2, Zabrze, Poland
- Hospital Juan Canalejo, As Xubias 84, La Coruna, Spain
- Inselspital - Universitätsspital Bern Postfach 33, Schweizer Herz-und Gefässzentrum Bern, Canton of Bern, Switzerland
- Papworth Hospital, Papworth Everard, Cambridge, United Kingdom

REFERENCES:
- [Derived] Crespo-Leiro MG, Stypmann J, Schulz U, Zuckermann A, Mohacsi P, Bara C, Ross H, Parameshwar J, Zakliczynski M, Fiocchi R, Hoefer D, Colvin M, Deng MC, Leprince P, Elashoff B, Yee JP, Vanhaecke J. Clinical usefulness of gene-expression profile to rule out acute rejection after heart transplantation: CARGO II. Eur Heart J. 2016 Sep 1;37(33):2591-601. doi: 10.1093/eurheartj/ehv682. Epub 2016 Jan 7. PMID 26746629
- [Derived] Crespo-Leiro MG, Stypmann J, Schulz U, Zuckermann A, Mohacsi P, Bara C, Ross H, Parameshwar J, Zakliczynski M, Fiocchi R, Hoefer D, Deng M, Leprince P, Hiller D, Eubank L, Deljkich E, Yee JP, Vanhaecke J. Performance of gene-expression profiling test score variability to predict future clinical events in heart transplant recipients. BMC Cardiovasc Disord. 2015 Oct 9;15:120. doi: 10.1186/s12872-015-0106-1. PMID 26452346
- [Derived] Crespo-Leiro MG, Zuckermann A, Bara C, Mohacsi P, Schulz U, Boyle A, Ross HJ, Parameshwar J, Zakliczynski M, Fiocchi R, Stypmann J, Hoefer D, Lehmkuhl H, Deng MC, Leprince P, Berry G, Marboe CC, Stewart S, Tazelaar HD, Baron HM, Coleman IC, Vanhaecke J. Concordance among pathologists in the second Cardiac Allograft Rejection Gene Expression Observational Study (CARGO II). Transplantation. 2012 Dec 15;94(11):1172-7. doi: 10.1097/TP.0b013e31826e19e2. PMID 23222738